CLINICAL TRIAL: NCT03307057
Title: Promoting Transactional Supports to Optimize Social Communication Outcomes for Infants and Their Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jennifer Stapel-Wax, Professor, Emory University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00098127; P50MH100029 (NIH)
Record Dates: First submitted 2017-10-06; First posted 2017-10-11 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Pediatrics; Behavioral Research
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: This study uses a 2-stage sequential multiple assignment randomized trial (SMART) design to develop an adaptive intervention. Participants will be randomized into one of two study arms at Stage 1 (6 months of age) and re-randomized into one of four arms for Stage 2 at 12 months of age. Certain study arms during Stage 2 will only be available for participants who are showing early signs of ASD.
Who Masked: Outcomes Assessor
Masking Description: The diagnosticians for all measures will be kept blind to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Social Communication Growth Charts (SCGC) in Stage 1 Plus SCGC in Stage 2 (Experimental): This arm includes infant participants who did not show early signs of ASD at 12 months of age, following stage 1.
  In stage 1, infants at 6 months of age with a sibling who is diagnosed with ASD, were randomized to receive the Social Communication Growth Charts (SCGC) intervention for 6 months.
  In stage 2, infants at 12 months of age who are not showing early signs of ASD were re-randomized to receive the Social Communication Growth Charts (SCGC) intervention from 12 to 21 months of age.
  Interventions: Behavioral: Social Communication Growth Charts (SCGC)
- Social Communication Growth Charts (SCGC) in Stage 1 Plus Usual Care in Stage 2 (Experimental): This arm includes participants who did not show early signs of ASD at 12 months of age, following stage 1.
  In stage 1, infants at 6 months of age with a sibling who is diagnosed with ASD were randomized to receive the Social Communication Growth Charts (SCGC) intervention for 6 months.
  In stage 2, infants at 12 months of age who are not showing early signs of ASD were re-randomized to receive usual care from 12 to 21 months of age.
  Interventions: Behavioral: Social Communication Growth Charts (SCGC); Behavioral: Usual Care
- SCGC in Stage 1 Plus Parent-Implemented (P-I) Condition in Stage 2 (Experimental): This arm includes infant participants who show early signs of ASD at 12 months of age, following stage 1.
  In stage 1, infants at 6 months of age with a sibling who is diagnosed with ASD, were randomized to receive the Social Communication Growth Charts (SCGC) intervention for 6 months.
  In stage 2, infants at 12 months of age showing early signs of ASD were randomized to receive a parent-implemented (P-I) condition of a naturalistic developmental behavioral intervention (NDBI) from 12 to 21 months of age.
  Interventions: Behavioral: Social Communication Growth Charts (SCGC); Behavioral: Parent-Implemented (P-I) Condition
- SCGC in Stage 1 Plus Clinician-Implemented (C-I) Condition in Stage 2 (Experimental): This arm includes infant participants who show early signs of ASD at 12 months of age, following stage 1.
  In stage 1, infants at 6 months of age with a sibling who is diagnosed with ASD, were randomized to receive the Social Communication Growth Charts (SCGC) intervention for 6 months.
  In stage 2, infants at 12 months of age showing early signs of ASD were randomized to receive a clinician-implemented (C-I) condition NDBI based on a hybrid model from 12 to 21 months of age.
  Interventions: Behavioral: Social Communication Growth Charts (SCGC); Behavioral: Clinician-Implemented (C-I) Condition
- Usual Care in Stage 1 Plus SCGC in Stage 2 (Experimental): This arm includes infant participants who did not show early signs of ASD at 12 months of age, following stage 1.
  In stage 1, infants at 6 months of age with a sibling who is diagnosed with ASD, were randomized to receive usual care for 6 months.
  In stage 2, infants at 12 months of age who are not showing early signs of ASD were re-randomized to receive the Social Communication Growth Charts (SCGC) intervention from 12 to 21 months of age.
  Interventions: Behavioral: Social Communication Growth Charts (SCGC); Behavioral: Usual Care
- Usual Care in Stage 1 Plus Usual Care in Stage 2 (Active Comparator): This arm includes infant participants who did not show early signs of ASD at 12 months of age, following stage 1.
  In stage 1, infants at 6 months of age with a sibling who is diagnosed with ASD, were randomized to receive usual care for 6 months.
  In stage 2, infants at 12 months of age who are not showing early signs of ASD were re-randomized to receive usual care from 12 to 21 months of age.
  Interventions: Behavioral: Usual Care
- Usual Care in Stage 1 Plus Parent-Implemented (P-I) Condition in Stage 2 (Experimental): This arm includes infant participants who show early signs of ASD at 12 months of age, following stage 1.
  In stage 1, infants at 6 months of age with a sibling who is diagnosed with ASD, were randomized to receive usual care for 6 months.
  In stage 2, infants at 12 months of age showing early signs of ASD were randomized to receive a parent-implemented (P-I) condition of a naturalistic developmental behavioral intervention (NDBI) from 12 to 21 months of age.
  Interventions: Behavioral: Parent-Implemented (P-I) Condition; Behavioral: Usual Care
- Usual Care in Stage 1 Plus Clinician-Implemented (C-I) Condition in Stage 2 (Experimental): This arm includes infant participants who show early signs of ASD at 12 months of age, following stage 1.
  In stage 1, infants at 6 months of age with a sibling who is diagnosed with ASD, were randomized to receive usual care for 6 months.
  In stage 2, infants at 12 months of age showing early signs of ASD were randomized to receive a clinician-implemented (C-I) condition NDBI based on a hybrid model from 12 to 21 months of age.
  Interventions: Behavioral: Clinician-Implemented (C-I) Condition; Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Social Communication Growth Charts (SCGC) — The Social Communication Growth Charts (SCGC) is a web-based tool that parents can access to teach them the social communication milestones that are developing from 6 to 24 months of age. The SCGC has an explore function with hundreds of video clips illustrating 80 social communication milestones and a support video that has narration explaining how the parent in the video is supporting the child's development. The SCGC also has a charting function that parents can use by answering questions about their child's social communication milestones and then view charts in 5 developmental domains. Parents in the SCGC condition are also invited to a bi-weekly online Guided Tour to join other parents in a group meeting, like a book club, as they go through the SCGC.
  Arms: SCGC in Stage 1 Plus Clinician-Implemented (C-I) Condition in Stage 2; SCGC in Stage 1 Plus Parent-Implemented (P-I) Condition in Stage 2; Social Communication Growth Charts (SCGC) in Stage 1 Plus SCGC in Stage 2; Social Communication Growth Charts (SCGC) in Stage 1 Plus Usual Care in Stage 2; Usual Care in Stage 1 Plus SCGC in Stage 2
Behavioral: Parent-Implemented (P-I) Condition — The Parent-Implemented (P-I) condition is based on the Early Social Interaction (ESI) model, which is an evidence-based parent-implemented intervention involving active and productive engagement for 5 hours per day, 5 days per week for toddlers with ASD. ESI teaches parents how to support their child's social communication, language, play and behaviors in everyday routines, activities, and places.
  Weekly home sessions with a family navigator include:
  1. developing the visit agenda
  2. intervention implementation including: guided/caregiver practice, feedback and problem solving
  3. planning for parent implementation between sessions
  Families can also access the Autism Navigator How-To Guide for Families (a self-guided, web-based course), the Online Guided Tour for the How-To Guide (an online group to engage families), and have the opportunity to interact with other families who suspect their child has autism through audio or video conferencing or typed chat.
  Arms: SCGC in Stage 1 Plus Parent-Implemented (P-I) Condition in Stage 2; Usual Care in Stage 1 Plus Parent-Implemented (P-I) Condition in Stage 2
Behavioral: Clinician-Implemented (C-I) Condition — The Clinician-Implemented (C-I) condition is based on the core principles of empirically-supported naturalistic developmental behavioral interventions (NDBI) for infants and toddlers with or at-risk for ASD, including Early Start Denver Model (ESDM), Project ImPACT (Improving Parents As Communication Teachers), Pivotal Response Treatment (PRT), and Early Social Interaction (ESI). The goal of C-I NDBI is to use naturalistic, developmental, and behavioral strategies with infants at-risk for ASD to improve social-communication, which includes eye contact, gesture use, intentional vocalizations, and language. Parents are not actively involved in C-I NDBI intervention sessions, though they may observe and the clinician will be given information about current social-communication targets.
  Arms: SCGC in Stage 1 Plus Clinician-Implemented (C-I) Condition in Stage 2; Usual Care in Stage 1 Plus Clinician-Implemented (C-I) Condition in Stage 2
Behavioral: Usual Care — Care as recommended and provided by the child's pediatrician or other health care providers in the community.
  Arms: Social Communication Growth Charts (SCGC) in Stage 1 Plus Usual Care in Stage 2; Usual Care in Stage 1 Plus Clinician-Implemented (C-I) Condition in Stage 2; Usual Care in Stage 1 Plus Parent-Implemented (P-I) Condition in Stage 2; Usual Care in Stage 1 Plus SCGC in Stage 2; Usual Care in Stage 1 Plus Usual Care in Stage 2

SUMMARY:
This early treatment project is designed to address two significant public health challenges - the need for validated, manualized, treatments for young children with Autism Spectrum Disorder (ASD) that are cost-efficient and feasible for community-based implementation, and the need to reduce the age of entry into early intervention to optimize outcomes. This study will use a 2-stage sequential multiple assignment randomized trial (SMART) design to develop an adaptive intervention by comparing individual and combined effects of preventative parent education and autism treatment starting in infancy. All parent-infant dyads from the pool of 250 high and low risk siblings in the Emory Autism Center of Excellence (ACE) will be invited at 6 months of age and randomly assigned at Stage 1 to the Social Communication Growth Charts (SCGC) that use an innovative web-based technology to teach parents early social communication milestones and how to support their child's development very early or Usual Care (UC), in order to compare the efficacy on developmental trajectories from 9 to 30 months. Families of children who show early signs of ASD at 12 months of age based on tailoring variables using parent report and observational measures will be re-randomized at Stage 2 to compare efficacy of a parent-implemented (P-I) condition of a naturalistic developmental behavioral intervention (NDBI) based on the Early Social Interaction (ESI)1 model to a clinician-implemented (C-I) condition of NDBI based on a hybrid model from 12 to 21 months of age. The investigators anticipate that 80 children will show early signs of ASD and that 56 families (70%) will agree to participate in the Stage 2 treatment. Growth trajectories of parent contingent responsiveness and child social communication will be collected longitudinally with repeated measures at 9, 12, 16, 21, and 30 months. Outcome measures of autism symptoms, developmental level, and adaptive behavior will be examined at 21 and 30 months to measure differential treatment effects.

DETAILED DESCRIPTION:
Most children with autism spectrum disorders (ASD) require special education at school age at staggering expenses to the educational system. The average annual cost for educating a child with ASD, based on the US Government Accountability Office, is $18,790, compared to $12,500 for the average special education student, and $6,556 for a regular education student. With effective early intervention (EI) services, the future is more promising. Through prior research, it is known that providing intervention early has a greater impact; between 60 and 90% of children in intensive early treatment programs beginning by age 3 can learn to talk compared to 50% without early treatment, and about half can make it into regular kindergarten, compared to 10% without early treatment. While there is a national priority for early intervention as evident in the mandate of Part C of the Individuals with Disabilities Education Act (IDEA), there is a need for research on effective and feasible early intervention programs for infants and toddlers with ASD.

The recommendations of the American Academy of Pediatrics to screen all children for ASD at 18-24 months of age makes the need for evidence-based interventions for toddlers with ASD even more pressing. Advances in research have documented that ASD can be diagnosed reliably by trained professionals at 18-24 months of age. And yet, the median age of diagnosis in the US is 4-5 years. Lower income, minority, and rural families receive a diagnosis up to a year and a half later, well beyond the opportunity for EI. Because the usual age of diagnosis of ASD is between 3 and 6 years of age, there is limited research on early intervention for infants and toddlers with ASD. Disparities in the age of detection of ASD delay the age of entry into intervention for children from underserved families. Compounding this problem, underserved families are underrepresented in intervention research, making them a critically important population to target in future research. It is vitally important to develop and document the effectiveness of interventions that could be implemented by public IDEA Part C service delivery program in community-base settings and that are feasible for low income and other underserved families.

The overarching goal of this treatment project is to document the efficacy of very early transactional supports that parents can learn to change developmental trajectories and optimize outcomes of their child using a 2-stage sequential multiple assignment randomized trial (SMART) design to develop an adaptive intervention. All parent-infant dyads in the Emory Autism Center of Excellence (ACE) will be invited at 6 months of age from the pool of 250 high and low risk siblings and will be randomly assigned at Stage 1 of this clinical trial. In Stage 1, parents of participating children are randomized to a group utilizing the Social Communication Growth Charts (SCGC), which use an innovative web-based technology to teach parents early social communication milestones and how to support their child's very early development, or Usual Care (UC). This first stage of the study will compare efficacy of the SCGC on parent contingent responsiveness and child developmental trajectories.

Participants will be re-randomized into one of four arms for Stage 2 when the children are 12 months of age. Families of children who do not show singes of ASD at 12 months of age will be re-randomized to SCGC or UC. Families of children who show early signs of ASD at 12 months of age will be re-randomized in Stage 2 to a parent-implemented (P-I) condition or a clinician-implemented (C-I) condition. The goal of Stage 2 of the study is to compare the efficacy of a parent-implemented (P-I) condition of a naturalistic developmental behavioral intervention (NDBI) based on the Early Social Interaction model, to a clinician-implemented (C-I) condition NDBI based on a hybrid model. Children will receive the Stage 2 intervention from 12 to 21 months of age.

Outcome measures of social communication, autism symptoms, social visual engagement, developmental level, and adaptive behavior will be gathered every 6 months from 6 to 30 months of age to measure treatment effects. Measures of parent transactional support and child active engagement will be collected quarterly from 9 to 30 months of age to examine growth trajectories during the Stage 1 and 2 conditions and at follow-up at 21 and 30 months after intervention. The expected impact of this study will have the following important implications: 1) maximize the use of technology to teach all parents how to support their infant's development early to optimize opportunities for learning and recognize as early as possible if their child is not meeting developmental milestones and may need intervention; 2) document improved outcomes for very young children with early signs of ASD receiving a manualized, evidence-based NDBI intervention that is cost-efficient and feasible for community-based implementation; and 3) substantiate that these adaptive interventions implemented by parents beginning at 6 months of age lead to better child outcomes, providing evidence that very early detection of autism is crucial to improve developmental outcomes.

ELIGIBILITY:
Inclusion Criteria for Stage 1:

* Have an ASD sibling who is in the Emory Autism Center of Excellence.

Inclusion Criteria for Stage 2:

* Nonresponse to Stage 1 intervention; a "nonresponder" is defined as infants who show early signs of autism and communication delay.
* Shows early signs of ASD, defined by a positive score on the Infant-Toddler Checklist (ITC) and at least two of the following autism screening tools: Early Screening for Autism and Communication Disorders (ESAC), Systematic Observation of Red Flags of ASD (SORF) Clinic, or SORF-Home.

Exclusion Criteria:

* Parent/caregiver declines to participate.

Ages: 6 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 269 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Measure of Active Engagement and Transactional Supports (MAETS) Score | 9, 12, 16, 21, and 30 months of age
  Parent contingent responsiveness will be assessed using the Transactional Support section of the Measure of Active Engagement and Transactional Supports (MAETS). This assessment will occur during home observation of everyday activities. This section includes 8 components: promoting participation and a productive role, providing structure to make activities predictable, using language that follows the child's focus of attention, promoting child initiations, providing a balance of communicative turns, supporting the development of child comprehension, providing verbal and nonverbal models, caregiver creates appropriate expectations and demands. Each component is scored on a 4 point scale where 0 = Absent, 1 = Emerging, 2 = Practicing, 3 = Mastery. Total scores range from 0 to 32 and lower scores indicate that the level of support is low.
  Families assigned to the Social Communication Growth Charts (SCGC) will be compared with families assigned to Usual Care (UC).
Communication and Symbolic Behavior Scales (CSBS) Score | 9, 12, 16, 21, and 30 months of age
  Change in social communication skills will be measured with the Communication and Symbolic Behavior Scales (CSBS) Behavior Sample. Interactions between the child and caregiver will be videotaped and later converted scores. The raw scores will be summed to form a social, speech, and symbolic composite.
  The social composite includes emotion and eye gaze, communication and gestures, and possible composite scores range from 0 to 64. The speech composite includes sounds and words, and possible composite scores range from 0 to 54. The symbolic composite includes understanding and object use, and possible scores for this composite range from 0 to 53. The total summed score for all three composites range from 0 to 171.
  Families assigned to the Social Communication Growth Charts (SCGC) will be compared with families assigned to Usual Care (UC).
Autism Diagnostic Observation Schedule Score | 9, 12, 16, 21, and 30 months of age
  Autism symptoms will be measured with the Autism Diagnostic Observation Schedule, Second Edition is the best gold standard diagnostic measure of ASD. The revised algorithms forming Social-Affect and Restricted Repetitive Behavior ratings of autism symptoms will be used. A total of score of 1 to 3 indicates no signs of autism, a score of 4 or 5 suggests that the child may have autism spectrum disorder, while a score of 6 to 10 is indicative of autism.
  Families assigned to the Social Communication Growth Charts (SCGC) will be compared with families assigned to Usual Care (UC).
Mullen Scales of Early Learning Score | 9, 12, 16, 21, and 30 months of age
  This study will use four scales of the Mullen Scales of Early Learning (MSEL) to measure developmental level. with separate scores for four cognitive scales that form an early learning composite. A nonverbal developmental quotient (DQ) based on age equivalent divided by chronological age multiplied by 100 will be calculated from the average of the Fine Motor and Visual Reception scales. A verbal DQ will be calculated from the Expressive Language and Receptive Language scales.
  Families assigned to the Social Communication Growth Charts (SCGC) will be compared with families assigned to Usual Care (UC).
Vineland-3 Adaptive Behavior Scales Score | 9, 12, 16, 21, and 30 months of age
  Adaptive Behavior will be measured with the Vineland-3 Adaptive Behavior Scales. The Vineland-3 provides a standard score in four domains of Communication, Daily Living Skills, Socialization, and Motor Skills, which yield an Adaptive Behavior Composite score. The normative mean score of the Adaptive Behavior Composite is 100 with a normative standard deviation of 15.
  Families assigned to the Social Communication Growth Charts (SCGC) will be compared with families assigned to Usual Care (UC).
Measure of Active Engagement and Transactional Supports (MAETS) in Parents of Children Showing Signs of ASD | 12 months of age to 21 months of age
  Parent contingent responsiveness will be assessed during home observation of everyday activities. Families who receive the P-I condition as the adaptive intervention will be compared with those receiving the C-I intervention.
Communication and Symbolic Behavior Scales (CSBS) Score in Children Showing Signs of ASD | 12 months of age to 21 months of age
  Change in social communication skills will be measured with the Communication and Symbolic Behavior Scales (CSBS) Behavior Sample. Interactions between the child and caregiver will be videotaped and later converted scores. The raw scores will be summed to form a social, speech, and symbolic composite.
  The social composite includes emotion and eye gaze, communication and gestures, and possible composite scores range from 0 to 64. The speech composite includes sounds and words, and possible composite scores range from 0 to 54. The symbolic composite includes understanding and object use, and possible scores for this composite range from 0 to 53. The total summed score for all three composites range from 0 to 171.
  Families who receive the P-I condition as the adaptive intervention will be compared with those receiving the C-I intervention.
Autism Diagnostic Observation Schedule Score in Children Showing Signs of ASD | 12 months of age to 21 months of age
  Autism symptoms will be measured with the Autism Diagnostic Observation Schedule, Second Edition is the best gold standard diagnostic measure of ASD. The revised algorithms forming Social-Affect and Restricted Repetitive Behavior ratings of autism symptoms will be used. A total of score of 1 to 3 indicates no signs of autism, a score of 4 or 5 suggests that the child may have autism spectrum disorder, while a score of 6 to 10 is indicative of autism.
  Families who receive the P-I condition as the adaptive intervention will be compared with those receiving the C-I intervention.
Mullen Scales of Early Learning Score in Children Showing Signs of ASD | 12 months of age to 21 months of age
  This study will use four scales of the Mullen Scales of Early Learning (MSEL) to measure developmental level. with separate scores for four cognitive scales that form an early learning composite. A nonverbal developmental quotient (DQ) based on age equivalent divided by chronological age multiplied by 100 will be calculated from the average of the Fine Motor and Visual Reception scales. A verbal DQ will be calculated from the Expressive Language and Receptive Language scales.
  Families who receive the P-I condition as the adaptive intervention will be compared with those receiving the C-I intervention.
Vineland-3 Adaptive Behavior Scales Score in Children Showing Signs of ASD | 12 months of age to 21 months of age
  Adaptive Behavior will be measured with the Vineland-3 Adaptive Behavior Scales. The Vineland-3 provides a standard score in four domains of Communication, Daily Living Skills, Socialization, and Motor Skills, which yield an Adaptive Behavior Composite score. The normative mean score of the Adaptive Behavior Composite is 100 with a normative standard deviation of 15.
  Families who receive the P-I condition as the adaptive intervention will be compared with those receiving the C-I intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Call, PhD, Principal Investigator — Emory University
Locations (1):
- Marcus Autism Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT03307057/ICF_000.pdf